CLINICAL TRIAL: NCT02978859
Title: A Phase II Trial of Sitravatinib (MGCD516), a Multi-receptor Tyrosine Kinase Inhibitor, in Advanced Liposarcoma and Other Soft Tissue Sarcomas
Brief Title: Sitravatinib in Advanced Liposarcoma and Other Soft Tissue Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ8661
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Liposarcoma; Metastatic Liposarcoma
Keywords: MGCD516; Sarcoma; Liposarcoma; Unresectable Liposarcoma; Metastatic Liposarcoma; Sitravatinib
MeSH Terms: conditions — Liposarcoma; Sarcoma | interventions — sitravatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MGCD516 (Experimental): Patients with locally advanced and unresectable or metastatic sarcoma will receive MGCD516 at the discretion of the principal investigator until disease progression, unacceptable toxicity or adverse event(s) or withdrawal of consent.
  Interventions: Drug: MGCD516

INTERVENTIONS:
Drug: MGCD516 — Administered at 150 mg orally, daily, in continuous 21 day cycles. An orally available, potent small molecular inhibitor of several related receptor tyrosine kinases.
  Other Names: Sitravatinib

SUMMARY:
The purpose of this study is to evaluate Sitravatinib, an oral small molecular receptor tyrosine kinase inhibitor, for the treatment of advanced liposarcoma.

DETAILED DESCRIPTION:
Sarcomas are a group of cancers which arise from connective tissue and bone, of which more than 50 subtypes exist. Approximately 12,000 people are diagnosed with sarcoma annually in the United States.

Liposarcoma is one of the more common types of soft tissue sarcoma. The primary treatment for liposarcoma is surgery when possible. When liposarcoma is not amenable to surgery, various systemic treatments, including chemotherapy, are used. However, the effectiveness of existing treatments for liposarcoma is limited.

Sitravatinib is an oral, targeted drug which inhibits receptor tyrosine kinases. Receptor tyrosine kinases are proteins on the surface of the liposarcoma cell which play a role in cancer growth. In laboratory work, Sitravatinib effectively suppressed the growth of liposarcoma models. The purpose of this study is to evaluate the safety and efficacy of Sitravatinib in patients with liposarcoma which cannot be removed by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1, histologically confirmed well-differentiated or de-differentiated liposarcoma. If stage 1 of the Simon II stage design fails to meet its endpoint for liposarcoma patients, an additional 16 patients will be enrolled, composed of 4 each of MPNST, synovial sarcoma, alveolar rhabdomyosarcoma and alveolar soft part sarcoma (otherwise, an additional 16 patients with well-differentiated or de-differentiated liposarcoma would be enrolled). Pathology review occurs at the center enrolling the patient on this trial.
* Disease must be locally advanced and unresectable or metastatic. Disease which may be resected but with an associated level of morbidity deemed unacceptable by the treating clinician is considered eligible.
* Patients must have measurable disease by RECIST criteria version 1.1.
* Patients must evidence of disease progression, either clinically or radiographically,within the 8 weeks prior to study enrollment, as determined by the principal investigator.
* Patients must have been treated with at least one prior systemic regimen for sarcoma. Adjuvant systemic therapy qualifies as prior therapy for the purposes of this study. There is no upper limit on previous lines of therapy received. A prior line of systemic therapy may include prior investigational agents received as part of other clinical studies.
* Patients must be age 18 years or older. Because no dosing or adverse event data are currently available for MGCD516 in patients less than 18 years of age, children are excluded from the present study, but will be eligible for future pediatric trials.
* Patients must demonstrate an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients must demonstrate normal organ and marrow function.
* Patients must demonstrate adequately controlled blood pressure at the time of study entry, as defined by a blood pressure ≤ 150/100 mmHg at study screening on at least one of two screenings conducted at least 24 hours apart. If blood pressure meets these guidelines on initial measurement, no subsequent measurement for screening is needed. Blood pressure may be assessed by automated or manual methods by an appropriately trained clinician or nurse.
* Patients must have normal left ventricular systolic function, as demonstrated by a transthoracic echocardiogram or multigated acquisition (MUGA) scan showing a normal left ventricular ejection fraction.
* Women of child-bearing potential and all men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients must not have received treatment with any chemotherapy, immunotherapy, radiotherapy or an investigational agent for malignancy within the 28 days preceding study registration. Patients may not have received treatment with nitrosureas or mitomycin within the 42 days prior to study registration. Patients may not have received treatment with a small molecule targeted agent (including off-label or investigational use) within 14 days preceding study registration, provided this represents at least 7 half-lives for that agent. Toxic effects from any prior therapy (except alopecia) must have resolved to grade 1 or less according to NCI CTCAE v4.0 or to the patient's baseline by the time of registration.
* Patients may not be receiving any other investigational agent for any purpose concurrently. Patients may not require ongoing treatment with (a) gastric pH modifying medications including proton pump inhibitors or H2 blockers (patients may switch to antacids), (b) medications which are known to be sensitive substrates or substrates with a narrow therapeutic index for the P-gp and breast cancer resistance protein (BCRP) transporters and/or (c) medications known to cause corrected QT Interval (QTc) prolongation with risk of Torasades. Please see Appendix 1 for a list of such prohibited concomitant medications at study entry.
* Patients with brain metastases which are symptomatic may not be enrolled. Those subjects with untreated brain metastases ≤ 1 cm may who are asymptomatic and for whom there are no plans for surgery, radiation or corticosteroid use may be considered eligible at the discretion of the principal investigator. Subjects with brain metastases that have been treated and are stable for at least 1 month are eligible if they are asymptomatic and not receiving corticosteroids.
* Patients may not have a history of allergic reaction or hypersensitivity to microcrystalline cellulose (Avicel PH302) or polysorbate 80 (Tween 80), which are components of the drug product MGCD516.
* Patients may not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, uncontrolled diabetes mellitus or uncontrolled psychiatric illness that would limit compliance with study requirements in the opinion of the principal investigator. Additionally, patients must be free of any impairment in the ability to swallow and absorb the oral study drug.
* Patients may not be pregnant or nursing. Pregnant women are excluded from this study because the teratogenic effects of MGCD516 have not been adequately studied. A negative pregnancy test must be documented 7 days or less prior to registration. Because there is an unknown but potential risk for adverse events to nursing infants secondary to treatment of the mother with MGCD516, breastfeeding must be discontinued prior to registration for this clinical trial.
* Patients may not have known HIV infection. HIV-positive patients on combination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Izar, MD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Massachussetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MGCD516
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MGCD516
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 62 [38 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 22
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 29
DDLPS [Count of Participants; unit: Participants] — Patients with dedifferentiated liposarcoma (DDLPS) at the start of the study
  Participants | 27
WDLPS [Count of Participants; unit: Participants] — Patients with well-differentiated liposarcoma (WDLPS) at the start of the study
  Participants | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Progression Free
Description: The number of patients alive and without evidence of disease progression per RECIST criteria v1.1 at the 12-week scan after starting treatment.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MGCD516
Number analyzed (Participants) | 29
Participants | 12

2. Secondary Outcome: Number of Participants Who Experienced a Treatment-related Adverse Event
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MGCD516
Number analyzed (Participants) | 29
Participants | 25

3. Secondary Outcome: Overall Response Rate (ORR) of MGCD516
Description: The ORR was defined as the number of patients having a best objective tumor status of complete or partial response per RECIST v1.1 criteria lasting at least 4 weeks divided by the number of evaluable patients.
Time Frame: Up to 33 months
Measure: Number; unit: participants
Arm/Group | MGCD516
Number analyzed (Participants) | 29
participants | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined from the date of enrollment to the date of progression or death, the last progression-free scan for patients who withdrew consent or had unexpected adverse events, or the last follow-up for patients who withdrew consent prior to the first scan, whichever occurred first.
  PFS and OS were estimated using the Kaplan-Meier method.
Time Frame: Up to 33 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MGCD516
Number analyzed (Participants) | 29
weeks | 11.7 [5.9 to 35.9]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined from the date of enrollment to the date of death or last follow-up, whichever occurred first.
  PFS and OS were estimated using the Kaplan-Meier method.
Time Frame: Up to 33 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MGCD516
Number analyzed (Participants) | 29
weeks | 31.7 [18.1 to 90.1]

ADVERSE EVENTS:
Time Frame: Up to 33 months
Arm/Group | MGCD516
All-Cause Mortality (participants affected / at risk) | 21/29
Serious Adverse Events (participants affected / at risk) | 12/29
Other Adverse Events (participants affected / at risk) | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MGCD516 (N=29)
Hypertension (Grade 3 and 4) (General disorders) | 7
Fatigue (Grade 3) (General disorders) | 2
Oral mucositis (Grade 3) (General disorders) | 1
Anemia (Grade 3) (Vascular disorders) | 1
Weight loss (Grade 3) (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MGCD516 (N=29)
Diarrhea (Gastrointestinal disorders) | 17
Hypertension (Grades 1 and 2) (General disorders) | 8
Fatigue (General disorders) | 11
Hoarseness (General disorders) | 12
Oral mucositis (Grades 1 and 2) (General disorders) | 8
Nausea (General disorders) | 9
Anorexia (General disorders) | 7
Constipation (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Anemia (Grade 1 and 2) (General disorders) | 4
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 5
Headache (General disorders) | 4
Weight loss (Grade 1 and 2) (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT02978859/Prot_SAP_000.pdf